CLINICAL TRIAL: NCT04894760
Title: Evaluation of a Rapid Diagnostic Test of SARS-COV-2 Carried Out in the Emergency Units of Reference Hospitals in Mexico and in Primary Care: Multi-center Study
Brief Title: Evaluation of a COVID-19 Rapid Diagnostic Test in ER Departments in Mexico: a Multi-center Study
Status: Completed | Type: Observational
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: Rapid Test COVID
Record Dates: First submitted 2021-04-12; First posted 2021-05-20 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: rapid test; diagnosis; antigen test
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasal swab sampling and Saliva testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Rapid Antigen Test (PanBio Ag test) — Rapid Antigen Test (PanBio Ag test)

SUMMARY:
An observational (cross-sectional) study in the emergency services of participating hospitals, receiving patients with COVID-19 and influenza, aiming to evaluate the diagnostic performance of the rapid antigen detection test for COVID-19 both in nasal sampling and saliva, in patients attending emergency services in the 2020-2021 winter season, performed on site, compared to the gold standard (RT-qPCR).

DETAILED DESCRIPTION:
This study aims to analyze the usefulness of rapid tests, especially: a) as a diagnostic test in people attending care for nonspecific, respiratory symptoms, in emergency services of referral hospitals b) as a diagnostic test in contacts of known patients. c) as a diagnostic test to differentiate influenza from COVID-19 in the circumstance of an overlap of both viruses in the community. d) In the 3 cases, the gold standard would be the RT-PCR test for influenza and for SARS-COV-2 performed in the usual laboratory following the officially approved technique in Mexico. If the test were in saliva, it would also be much more accepted and could come close to performing a test at home that would greatly facilitate the diagnosis. So it is important to see the performance of a saliva test.

As an observational (cross-sectional) study in the emergency services of participating hospitals, receiving patients with COVID-19 and influenza, aiming to evaluate the diagnostic performance of the rapid antigen detection test for COVID-19 both in nasal sampling and saliva, in patients attending emergency services in the 2020-2021 winter season, performed on site, compared to the gold standard (RT-qPCR).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Signed Informed consent
* Emergency room visit or screening site with respiratory symptoms consistent with COVID-19 / influenza.

Exclusion Criteria:

* Positive pregnancy test
* Lactation
* Decision of the responsible physician to remove patient from the study.
* Transfer of the patient to another hospital unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that arrive to the ER department of each reference center.
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | At 24 hours
  Compared with gold standard RT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, "Ismael Cosío Villegas", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
No plan yet